CLINICAL TRIAL: NCT00896636
Title: Gene Methylation and Estradiol Levels in Random FNA Samples as Biomarkers for Breast Cancer Risk
Brief Title: Study of Breast Tissue in Women Not Previously Diagnosed With Breast Cancer Who Are Undergoing Fine Needle Aspiration
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Northwestern University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: NU 08B2; P30CA060553 (NIH); NU-08B2; NU-IRB-STU00003136
Record Dates: First submitted 2009-05-09; First posted 2009-05-12 (Estimated); Last update posted 2020-08-31 (Actual); Status verified 2020-08

CONDITIONS: Breast Cancer; Healthy, no Evidence of Disease
Keywords: breast cancer; healthy, no evidence of disease
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Breast tissue random fine needle aspiration (rFNA) samples will be collected and levels of methylation and hormones will be measured in each.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Luteal: Pre-menopausal women who undergo rFNA procedure during the luteal phase of their menstrual cycle.
  Interventions: Procedure: Random fine need aspiration (rFNA); Other: Mammogram
- Follicular: Pre-menopausal women who undergo rFNA procedure during the follicular phase of their menstrual cycle.
  Interventions: Procedure: Random fine need aspiration (rFNA); Other: Mammogram
- Menopause: Women who have entered menopause.
  Interventions: Procedure: Random fine need aspiration (rFNA); Other: Mammogram

INTERVENTIONS:
Procedure: Random fine need aspiration (rFNA) — Deep infiltration into the tissue of each breast with up to a 21 gauge needle attached to a syringe with about 4-5 passes at each location (up to 8-10 passes per breast) under local anesthesia (lidocaine).
Other: Mammogram — Standard mammography of both breasts to obtain images for breast density measurement.

SUMMARY:
RATIONALE: Studying samples of blood and breast tissue from healthy women in the laboratory may help doctors learn more about changes that occur in DNA and identify biomarkers related to breast cancer risk.

PURPOSE: This research study is looking at breast tissue in women not previously diagnosed with breast cancer who are undergoing fine-needle aspiration.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine if breast tissue DNA methylation profile and hormone concentration change across follicular and luteal phase, or across menopause, in random fine needle aspiration samples of women with no prior diagnosis or treatment for breast cancer.
* To determine if DNA methylation profile and breast hormone levels correlate with mammographic density, cytomorphology, or Gail risk estimates.
* To develop a high throughput commercial assay for DNA methylation profiling for assessing breast cancer risk.
* To develop a highly sensitive, specific, and novel nanoassay for estradiol and progesterone.

OUTLINE: This is a multicenter study.

Premenopausal women are stratified by menstrual cycle phase (mid-follicular [day 5-10] vs mid-luteal [day 20-25]), based on an adjusted 28-day cycle.

Patients undergo breast density measurement by digital mammography. Blood samples are obtained and analyzed for estradiol, progesterone, and follicle-stimulating hormone measurements, to define menstrual/menopausal status, and for DNA extraction. Patients also undergo random fine needle aspiration. Biopsy material from aspiration is analyzed for cytomorphology, steroid radioimmunoassay (RIA), steroid nanoassay, and DNA methylation studies (via polymerase chain reaction). The aspiration samples are also analyzed for estradiol and progesterone levels using high-pressure liquid chromatography and RIA.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Women meeting one of the following requirements:

  * Regularly cycling premenopausal women under 45 years of age
  * Perimenopausal women 45-55 years of age who have had ≥ two periods in the past 6 months
  * Postmenopausal women under 60 years of age (no menstrual period for 12 months and follicle-stimulating hormone (FSH) levels > 25 IU/dL)
* No history of breast cancer diagnosis or prior treatment for breast cancer
* Negative breast evaluation within the past 3 months

PATIENT CHARACTERISTICS:

* See Disease Characteristics

PRIOR CONCURRENT THERAPY:

* No concurrent oral contraceptives
* At least 2 weeks since prior aspirin, non-steroidal anti-inflammatory drugs, and vitamin E

Ages: 35 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Women coming in for screening mammography, for diagnostic imaging, for evaluation of benign breast problems, and for breast cancer risk evaluation who have no history of breast cancer.
Sampling Method: Non-Probability Sample
Enrollment: 385 (Actual)
Dates: Start 2009-02-20 (Actual); Primary Completion 2013-01-18 (Actual); Study Completion 2022-01 (Estimated)

PRIMARY OUTCOMES:
Differences in DNA methylation profiles between women in different menstrual stages | One time rFNA procedure to collect samples.
Differences in DNA methylation profiles between women in different menstrual stages | One time rFNA procedure to collect samples
Correlation between DNA methylation profiles and mammographic density, cytomorphology, or Gail risk estimate | One time rFNA procedure to collect sample to compare with baseline mammogram and risk info.

CONTACTS AND LOCATIONS:
Overall Officials: Seema A. Khan, MD, Principal Investigator — Robert H. Lurie Cancer Center
Locations (1):
- Robert H. Lurie Comprehensive Cancer Center at Northwestern University, Chicago, Illinois, United States